CLINICAL TRIAL: NCT00593489
Title: Advancing INSIGHT Methods in General Practice
Brief Title: Advancing Insulin Prescribing in General Practice
Acronym: AIM@GP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Stewart Harris, Professor, Family Medicine, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R-06-851; Lantu-L-01961 (Other Grant/Funding Number: Sanofi-aventis)
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus
Keywords: Insulin; Diabetes Mellitus; Practice Behaviour; Preceptor; Pharmacy
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Pharmacists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Basal Insulin Initiation Strategy (Experimental): Basal Insulin Initiation Strategy which includes:
  1. support by community pharmacist
  2. support by diabetes specialist
  Interventions: Other: Basal Insulin Initiation Strategy
- Usual Practice (No Intervention): The physicians randomized to this group proceeded with their usual practice

INTERVENTIONS:
Other: Basal Insulin Initiation Strategy — This multifaceted intervention consists of (1) Diabetes Specialist Consultation Support which entails specialists and educators providing consultation for insulin initiation and titration for the 12 months following the Workshop. Support will consist of prearranged and scheduled communications to review and advise for the first 2 months and will continue on an ad hoc basis for the remaining 10 months, with communication initiated by the physician (2)Community Pharmacy Insulin Initiation consists of trained community pharmacists providing patient education insulin initiation. Education will consist of one individual teaching session, one hour in duration, to review the insulin prescription protocol, insulin injection method, management of hypoglycemia, and self-monitoring of blood glucose.
  Other Names: Support by Specialist and Pharmacist
  Arms: Basal Insulin Initiation Strategy

SUMMARY:
Family Physicians, the subjects of this trial are reluctant to initiate insulin in patients with type 2 diabetes due to a lack of familiarity and comfort with this clinical strategy. This study will test the effectiveness of diabetes specialist consultation support, and community pharmacy insulin initiation support on the insulin prescribing behaviour of family physicians across Canada.

DETAILED DESCRIPTION:
The 2003 Canadian Diabetes Association clinical practice guidelines recommend early and sustained glycemic control targeting an glycosylated hemoglobin (A1C) < 7%. The guideline target however is not achieved in 50% of patients with type 2 diabetes in the Canadian family practice setting. Family physicians are not comfortable initiating and managing insulin for their patients the Diabetes in Canada Evaluation (DICE) study found that only 12% of the 2473 patients audited were prescribed insulin; 6% insulin alone and 6% in combination. Harris et. al. found 20% of patients prescribed insulin, 15% insulin alone and 5% in combination. A strategy to increase physicians' knowledge, skill and comfort with insulin prescription is needed to better achieve glycemic control for patients with type 2 diabetes in Canada.

Purpose - The purpose of AIM@GP is to increase family physicians clinical experience and comfort with insulin prescription and better achieve glycemic control for patients with type 2 diabetes in Canada.

Primary Objective - To determine the effectiveness of a Basal Insulin Initiation strategy on family physician insulin prescribing behaviour. The strategy, using a multifaceted behaviour facilitation approach, includes diabetes specialist consultation support, and community pharmacy insulin initiation support.

Study Design - The study design is a stratified, parallel group, randomized control effectiveness study. All physicians will attend an insulin education workshop where they will receive a Diabetes Practice Profile and randomly allocated in a 1:1 manner into the intervention or control group.

ELIGIBILITY:
Inclusion Criteria:

* Full time family physicians (FP) >25 hours per week in office
* Ability to generate a listing of patients with type 2 diabetes (T2DM) from their practice or billing records.
* Generation of a practice list of patients with T2DM
* A minimum of 50 patients with type 2 diabetes in their practice.
* Support the generation of a Diabetes Practice Profile prior to the deadline established
* A minimum of 6 insulin-eligible patients
* Attendance at the scheduled Workshop (if unable to attend the Workshop must be available to be educated and trained by diabetes nurse educator(DNE) using a Workshop DVD)

Exclusion Criteria:

* FP does not attend Workshop or complete educational training using Workshop DVD with DNE guidance
* FPs who anticipate retiring within the post-intervention period, moving their practice to another city, or having locum coverage of their practice for more than 4 weeks during the post-intervention period
* FPs currently participating in a diabetes behaviour-change intervention trial
* FPs working in an academic environment
* FPs unlikely to comply with protocol, (uncooperative attitude, unlikelihood of completing the study).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2006-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stewart B. Harris, MD MPH FCFP, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Lawson Health Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers

REFERENCES:
- [Background] Harris SB, Stewart M, Brown JB, Wetmore S, Faulds C, Webster-Bogaert S, Porter S. Type 2 diabetes in family practice. Room for improvement. Can Fam Physician. 2003 Jun;49:778-85. PMID 12836867
- [Background] Harris, Stewart B., Ekoe, J. M., and Webster-Bogaert, M. S. The Diabetes in Canada Evaluation (DICE) Study: Are Primary Care Physicians Achieving Target A1c? Diabetes 52(Supplement 1), A499. 2003.
- [Derived] Harris SB, Gerstein HC, Yale JF, Berard L, Stewart J, Webster-Bogaert S, Tompkins JW. Can community retail pharmacist and diabetes expert support facilitate insulin initiation by family physicians? Results of the AIM@GP randomized controlled trial. BMC Health Serv Res. 2013 Feb 21;13:71. doi: 10.1186/1472-6963-13-71. PMID 23433347

RESULTS

PARTICIPANT FLOW:
Groups:
- Basal Insulin Strategy: Basal Insulin Strategy
  1. Support by community pharmacist
  2. Support by diabetes specialist
- Usual Care: usual care - no intervention
Period: Allocation
Arm/Group | Basal Insulin Strategy | Usual Care
Started | 75 (allocated to intervention group to receive the intervention) | 79 (allocated to usual care group)
Completed | 73 | 78
Not Completed | 2 | 1
Not completed — did not attend workshop; allocation not | 2 | 1
Period: Analysis
Arm/Group | Basal Insulin Strategy | Usual Care
Started | 73 (physician withdrawal (N=3) primary outcome set to 0) | 78 (physician withdrawal (N=3) primary outcome set to 0)
Completed | 73 | 78
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of physicians randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Basal Insulin Strategy | Usual Care | Total
Number analyzed (Participants) | 75 | 79 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (8.81) | 48.2 (9.06) | 49.6 (9.12)
Sex: Female, Male [Count of Participants; unit: Participants] — The gender of the physician was ascertained by questionnaire and by direct communication
  Participants
    Female | 22 | 20 | 42
    Male | 53 | 59 | 112

OUTCOME MEASURES:

1. Primary Outcome: Insulin Prescription Rate - the Number of Insulin-eligible Patients Per 12 Months Who Are Prescribed Insulin in Each Family Physician (FP) Practice
Description: Insulin Prescription Rate (IPR) - the number of insulin-eligible patients per 12 months who are prescribed insulin in each family physician (FP) practice (Number of patients per year per FP). The IPR was analyzed using Poisson regression with the intervention group as a class effect and the mean HbA1c at baseline as a covariate.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: patients per year
Arm/Group | Basal Insulin Strategy | Usual Care
Number analyzed (Participants) | 73 | 78
patients per year | 2.28 (0.27) | 2.29 (0.25)
Statistical Analysis 1: Comparison: Basal Insulin Strategy vs Usual Care; The IPR was analyzed using Poisson regression with the intervention group as a class effect and the mean HbA1c at baseline as a covariate; Test type: Superiority; p = 0.96, Poisson Regression; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.8 to 1.24]

2. Secondary Outcome: Mean A1C of Insulin-eligible Patient Per Family Physician Post-Workshop
Description: mean A1C of insulin-eligible patient per family physician participant during the post-Workshop period
Time Frame: 15 months
Population: The analysis of secondary data was based on available data
Measure: Mean (Standard Deviation); unit: Mean % glycolyslated hemoglobin per FP
Arm/Group | Basal Insulin Strategy | Usual Care
Number analyzed (Participants) | 73 | 76
Mean % glycolyslated hemoglobin per FP
  Workshop | 7.12 (0.42) | 7.20 (0.52)
  End of Study | 7.09 (0.41) | 7.15 (0.51)

3. Secondary Outcome: Mean Fasting Blood Glucose of Insulin-eligible Patients
Description: mean fasting blood glucose (FBG) of insulin-eligible patient per family physician post-Workshop
Time Frame: 15 months
Population: The analysis of secondary data was based on available data
Measure: Mean (Standard Deviation); unit: mean mmol/L per physician
Arm/Group | Basal Insulin Strategy | Usual Care
Number analyzed (Participants) | 71 | 70
mean mmol/L per physician
  Workshop | 7.86 (0.67) | 7.89 (0.69)
  End of Study | 7.78 (0.68) | 7.82 (0.68)

4. Secondary Outcome: Percent of Insulin-eligible Patients With Intensification of Diabetes Management Per FP Post - Workshop
Description: Percent of insulin-eligible patients with intensification of diabetes management (increase dose of oral anti-diabetes drug (OAD) or insulin, OAD score, the addition of insulin) per FP post - Workshop
Time Frame: 12 months
Population: The analysis of secondary data was based on available data
Measure: Mean (Standard Deviation); unit: % of pts with intensification per FP
Arm/Group | Basal Insulin Strategy | Usual Care
Number analyzed (Participants) | 73 | 76
% of pts with intensification per FP | 31.59 (14.17) | 32.80 (14.91)

5. Secondary Outcome: Percentage of Patients at Target (A1C ≤ 7.0%) Per FP
Description: Percentage of patients at target (A1C ≤ 7.0%) per FP at time of the Workshop and post - Workshop
Time Frame: 15 months
Population: The analysis of secondary data was based on available data
Measure: Mean (Standard Deviation); unit: percentage of patients per physician
Arm/Group | Basal Insulin Strategy | Usual Care
Number analyzed (Participants) | 73 | 76
percentage of patients per physician
  Workshop | 58.4 (16.20) | 55.95 (15.65)
  End of Study | 58.68 (15.40) | 57.58 (16.12)

6. Secondary Outcome: Percent of Patients at Target (A1C ≤ 6.5%) Per FP
Description: Percent of patients at target (A1C ≤ 6.5%) per FP at time of the Workshop and post - Workshop
Time Frame: 15 months
Population: The analysis of secondary data was based on available data
Measure: Mean (Standard Deviation); unit: percent of patients per physician
Arm/Group | Basal Insulin Strategy | Usual Care
Number analyzed (Participants) | 70 | 73
percent of patients per physician
  At time of Workshop | 36.76 (14.95) | 36.62 (12.55)
  15 months post Workshop | 36.13 (15.06) | 36.61 (14.28)

7. Secondary Outcome: Change in "Insulin Prescription Rate"
Description: change in "Insulin Prescription Rate" from baseline prior to the Workshop to 12 months post - Workshop
Time Frame: 12 months
Population: In an updated version of the statistical analysis plan this variable was not calculated from the data set and not included in the analysis
Groups:
- Basal Insulin Initiation Strategy: Basal Insulin Initiation Strategy which includes:
  1. support by community pharmacist
  2. support by diabetes specialist
  Basal Insulin Initiation Strategy: This multifaceted intervention consists of (1) Diabetes Specialist Consultation Support which entails specialists and educators providing consultation for insulin initiation and titration for the 12 months following the Workshop. Support will consist of prearranged and scheduled communications to review and advise for the first 2 months and will continue on an ad hoc basis for the remaining 10 months, with communication initiated by the physician (2)Community Pharmacy Insulin Initiation consists of trained community pharmacists providing patient education insulin initiation. Education will consist of one individual teaching session, one hour in duration, to review the insulin prescription protocol, insulin injection method, management of hypoglycemia, and self-monitoring of blood glucose.
Arm/Group | Basal Insulin Initiation Strategy | Usual Practice
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Glycemic Control (A1C) at Insulin Initiation, 3 and 6 Months Post Initiation
Description: Glycemic control (A1C) at insulin initiation, 3 months post initiation and 6 months post initiation for those prescribed insulin per family physician
Time Frame: 15 months
Population: The analysis of secondary data was based on available data
Measure: Mean (Standard Deviation); unit: Mean % glycosylated hemoglobin per FP
Arm/Group | Basal Insulin Initiation Strategy | Usual Practice
Number analyzed (Participants) | 39 | 44
Mean % glycosylated hemoglobin per FP
  Initiation | 8.82 (1.098) | 9.37 (1.354)
  3 months post initiation | 8.32 (1.24) | 9.05 (1.344)
  6 months post initiation | 7.97 (1.003) | 8.57 (1.382)

9. Secondary Outcome: Physician Score for Knowledge of Insulin Initiation & Titration
Description: physician score for knowledge of insulin initiation & titration minimum score of 0 maximum score of 17. The greater the score the greater the knowledge.
Time Frame: 12 months
Population: The analysis of secondary data was based on available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Basal Insulin Initiation Strategy | Usual Practice
Number analyzed (Participants) | 59 | 59
units on a scale
  Pre-Workshop | 15.5 (2.2) | 15.5 (2.5)
  Post-Workshop | 16.3 (1.9) | 16.9 (1.9)

10. Secondary Outcome: Physician Score for Attitude Towards Insulin Initiation & Titration
Description: physician score for attitude towards insulin initiation & titration The minimum score is 11 and the maximum is 55 with a lower score indicating the ideal attitude.
Time Frame: 12 months
Population: The analysis of secondary data was based on available data"
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Basal Insulin Initiation Strategy | Usual Practice
Number analyzed (Participants) | 59 | 59
units on a scale
  Pre-Workshop | 28.9 (4.9) | 29.7 (5.3)
  Post-Workshop | 26.1 (4.1) | 27.3 (5.3)

11. Secondary Outcome: Physician Score for Self-efficacy of Insulin Initiation & Titration
Description: physician score for self-efficacy of insulin initiation & titration where the minimum value was 10 and the maximum was 50. A value of 50 indicated complete self efficacy to initiate and titrate insulin
Time Frame: 12 months
Population: The analysis of secondary data was based on available data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Basal Insulin Initiation Strategy | Usual Practice
Number analyzed (Participants) | 59 | 59
score on a scale
  Pre Workshop | 35.8 (4.67) | 35.7 (3.94)
  Post Workshop | 40.6 (3.73) | 39.6 (4.0)

ADVERSE EVENTS:
Description: ClinicalTrials.gov definition of adverse event (AE) is not applicable as the intervention was directed towards changing physician behaviour.
  Non-systematic Assessment was chosen Collection Approach for Table Default because it was a required field
  AE information was not gathered so zeros were entered for Numbers of Patients Affected and Numbers of Participants at Risk of AE. Zero was entered into Frequency Threshold for Reporting Other Adverse Events because it required a response.
Groups:
- Usual Care: usual care used as the control
Arm/Group | Basal Insulin Strategy | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The estimated sample size of 89 physicians/group was not achieved hence the final results may have been under-powered

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No